CLINICAL TRIAL: NCT00844649
Title: A Randomized Phase III Study of Weekly ABI-007 Plus Gemcitabine Versus Gemcitabine Alone in Patients With Metastatic Adenocarcinoma of the Pancreas
Brief Title: Phase III Study of ABI-007(Albumin-bound Paclitaxel) Plus Gemcitabine Versus Gemcitabine in Metastatic Adenocarcinoma of the Pancreas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA046
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albumin-bound paclitaxel (ABI-007)/Gemcitabine (Experimental): ABI-007 125 mg/m2 administered in combination with gemcitabine 1000 mg/m2 weekly for 3 weeks followed by one week of rest.
  Interventions: Drug: Albumin-bound paclitaxel (ABI-007); Drug: Gemcitabine
- Gemcitabine (Active Comparator): Gemcitabine, 1000 mg/m2 administered weekly for 7 weeks followed by a week of rest (Cycle 1), followed by cycles of weekly administration for 3 weeks followed by a week of rest (Cycle 2 onward).
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Albumin-bound paclitaxel (ABI-007) — ABI-007 125 mg/m^2 administered by intravenous infusion
  Other Names: Abraxane
  Arms: Albumin-bound paclitaxel (ABI-007)/Gemcitabine
Drug: Gemcitabine — Gemcitabine, 1000 mg/m2 administered weekly for 7 weeks, Day 1 through Day 43 followed by a week of rest (Cycle 1), followed by cycles of weekly administration for 3 weeks, Days 1, 8, and 15 followed by a week of rest (Cycle 2 onward).
  Other Names: Gemzar

SUMMARY:
Phase III Metastatic Pancreatic Cancer

DETAILED DESCRIPTION:
A Phase III, open-label randomized, multicenter trial to compare ABI-007(Albumin-bound Paclitaxel)in combination with gemcitabine administered weekly to standard treatment (gemcitabine monotherapy) with respect to overall survival, objective tumor response rate and Progression Free Survival (PFS) in patients diagnosed with metastatic adenocarcinoma of the pancreas.

ELIGIBILITY:
Inclusion Criteria

A participant will be eligible for inclusion in this study only if all of the following criteria are met:

1. Participant has definitive histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas. The definitive diagnosis of metastatic pancreatic adenocarcinoma will be made by integrating the histopathological data within the context of the clinical and radiographic data. Participants with islet cell neoplasms are excluded.
2. Initial diagnosis of metastatic disease must have occurred ≤6 weeks prior to randomization in the study.
3. Patient has one or more metastatic tumors measurable by Computed Tomography (CT) scan or Magnetic resonance imaging (MRI), if patient is allergic to CT contrast media).
4. Male or non-pregnant and non-lactating female, and ≥ 18 years of age. If a female patient is of child-bearing potential, as evidenced by regular menstrual periods, she must have a negative serum pregnancy test Beta-Human Chorionic Gonadotropin (β-hCG) documented 72 hours prior to the first administration of study drug.

   If sexually active, the patient must agree to use contraception considered adequate and appropriate by the Investigator during the period of administration of study drug. In addition, male and female patients must utilize contraception after the end of treatment as recommended in the product's Summary of Product Characteristics or Prescribing Information provided in the study manual.
5. Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatment with 5-Fluorouracil (5-FU) or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present. Patients having received cytotoxic doses of gemcitabine or any other chemotherapy in the adjuvant setting are not eligible for this study.
6. Patient has adequate biological parameters as demonstrated by the following blood counts at Baseline (obtained ≤14 days prior to randomization):

   Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; Platelet count ≥ 100,000/mm^3 (100 × 10^9/L); Hemoglobin (Hgb) ≥ 9 g/dL.
7. Patient has the following blood chemistry levels at Baseline (obtained ≤14 days prior to randomization):

   Aspartate Transaminase (AST), Serum Glutamic-Oxaloacetic Transaminase (SGOT), Alanine Transaminase ( ALT) Serum Glutamic-Pyruvic Transaminase (SGPT) ≤ 2.5 × upper limit of normal range (ULN), unless liver metastases are clearly present, then ≤ 5 × ULN is allowed Total bilirubin ≤ ULN Serum creatinine within normal limits or calculated clearance ≥ 60 mL/min/1.73 m^2 for patients with serum creatinine levels above or below the institutional normal value. If using creatinine clearance, actual body weight should be used for calculating creatinine clearance (e.g., using the Cockroft-Gault formula). For patients with a Body Mass Index (BMI) >30 kg/m^2, lean body weight should be used instead.
8. Patient has acceptable coagulation studies (obtained ≤14 days prior to randomization) as demonstrated by prothrombin time (PT) and partial thromboplastin time (PTT) within normal limits (± 15%).
9. Patient has no clinically significant abnormalities in urinalysis results (obtained ≤14 days prior to randomization).
10. Patient has a Karnofsky performance status (KPS) ≥ 70. Two observers will be required to assess KPS. If discrepant, the one with the lowest assessment will be considered true.
11. Patients should be asymptomatic for jaundice prior to Day 1. Significant or symptomatic amounts of ascites should be drained prior to Day 1. Pain symptoms should be stable and should not require modifications in analgesic management prior to Day 1.
12. Patient has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent Form (ICF) prior to participation in any study-related activities.

Exclusion Criteria

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

1. Patient has known brain metastases, unless previously treated and well-controlled for at least 3 months (defined as clinically stable, no edema, no steroids and stable in 2 scans at least 4 weeks apart).
2. Patient has only locally advanced disease.
3. Patient has experienced a ≥10% decrease in KPS between baseline visit and within 72 hours prior to randomization.
4. Patient has a ≥20% decrease in serum albumin level between baseline visit and within 72 hours prior to randomization.
5. History of malignancy in the last 5 years. Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Patients with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 5 years.
6. Patient uses Coumadin.
7. Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
8. Patient has known historical or active infection with Human Immunodeficiency Virus (HIV), hepatitis B, or hepatitis C.
9. Patient has undergone major surgery, other than diagnostic surgery (i.e.--surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
10. Patient has a history of allergy or hypersensitivity to any of the study drugs or any of their excipients, or the patient exhibits any of the events outlined in the Contraindications or Special Warnings and Precautions sections of the product or comparator Summary of Product Characteristics (SmPC) or Prescribing Information.
11. History of connective tissue disorders (e.g., lupus, scleroderma, arteritis nodosa).
12. Patients with a history of interstitial lung disease.
13. History of chronic leukemias (e.g., chronic lymphocytic leukemia).
14. Patients with high cardiovascular risk, including, but not limited to, recent coronary stenting or myocardial infarction in the past year.
15. History of Peripheral Artery Disease (e.g,. claudication, Leo Buerger's disease).
16. Patient has serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the patient's safety or the study data integrity.
17. Patient is enrolled in any other clinical protocol or investigational trial.
18. Patient is unwilling or unable to comply with study procedures, or is planning to take vacation for 7 or more consecutive days during the course of the study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 861 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2012-09-17 (Actual); Study Completion 2013-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Von Hoff, MD, Principal Investigator — Scottsdale Clinical Research Institute
Locations (193):
- United States (90):
  - UAB Comprenhensive Cancer Center at University of Alabama, Birmingham, Alabama
  - Clearview Cancer Institute Oncology Specialities, P.C., Huntsville, Alabama
  - TGEN Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - Mayo Clinic-Scottsdale, Scottsdale, Arizona
  - Northern Arizona Hematology and Oncology Associates-AOA, Sedona, Arizona
  - Arizona Cancer Center, University of Arizona, Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope, Duarte, California
  - Pacific Shores Medical Group, Long Beach, California
  - UCLA, Los Angeles, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - University Cancer Institute, LLC, Boynton Beach, Florida
  - Collaborative Research Group, Boynton Beach, Florida
  - FL Cancer Specialist, Fort Myers, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Lake County Oncology and Hematology, Tavares, Florida
  - Phoebe Putney Cancer Center, Albany, Georgia
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Piedmont Hospital Research Institute, Atlanta, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Atlanta Cancer Care, Atlanta, Georgia
  - Cancer Care & Hemaotology Specialists of Chicagoland, Arlington Heights, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Orchard Research, Skokie, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Hutchinson Clinic, PA, Hutchinson, Kansas
  - Owsley Brown Frazier Cancer Center, Louisville, Kentucky
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Mercy Hospital Portland, ME, Portland, Maine
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - Sidney Kimmel Comphrensive Cancer Center, John Hopkins University, Baltimore, Maryland
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - Cancer Center of Excellence/University of MA Medical School, Worcester, Massachusetts
  - St. Mary's/ Duluth Clinic, Duluth, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota
  - St. John's Medical Research Institute, Springfield, Missouri
  - Saint Louis University, St Louis, Missouri
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Hem Onc Associates-NM, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - New York Oncology Hematology PC, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Arena Oncology Associates, PC, Lake Success, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Piedmont Hematology Oncology, Winston-Salem, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Mid Ohio Oncology/Hematology Inc, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Cancer Centers of SW OK, Lawton, Oklahoma
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Mercy Physicians of Oklahoma, Oklahoma City, Oklahoma
  - Cancer Care Associates- Tulsa, Tulsa, Oklahoma
  - St. Mary Medical Center Hem-Onc Group, PC, Langhorne, Pennsylvania
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Medical City Dallas-US Oncology, Dallas, Texas
  - Texas Oncology, PA, Dallas, Texas
  - Texas Oncology, PA/ Methodist Charlton Cancer Center, Dallas, Texas
  - Texas Oncology Laboratories, Fort Worth, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - The University of Texas Medical School at Houston, Houston, Texas
  - Texas Oncology- Plano East, Plano, Texas
  - Texas Oncology, PA, Round Rock, Texas
  - Texas Oncology-Round Rock, Round Rock, Texas
  - South Texas Oncology and Hematology, P.A, San Antonio, Texas
  - Texas Oncology, PA, Wichita Falls, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fairfax-Northern Virginia Hematology-Oncology, P.C., Fairfax, Virginia
  - Virginia Cancer Specialist, PC, Fairfax, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Health Services, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Evergreen Hematology & Oncology, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (21):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Macarthur Cancer Therapy Center, Campbelltown, New South Wales
  - Concord Hospital, Concord, New South Wales
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Newcastle Hospital, Waratah, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Haemotology & Oncology Australasia (HOCA), Milton, Queensland
  - Haematology Oncology Clinics of Australasia-Gold Coast, Milton, Queensland
  - Adelaide Cancer Centre (T/A Ashford Cancer Ctr), Ashford, South Australia
  - Flinders Medical Center, Bedford Park, South Australia
  - Calvary North Adelaide Hospital, North Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Medical Oncology Unit, Bendigo Health, Bendigo, Victoria
  - Monash Medical Centre, East Bentleigh, Victoria
  - Western Hospital, Footscray, Victoria
  - Peninsula Oncology Centre, Frankston, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Perth, Western Australia
- Austria (4):
  - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - Landesklinikum St. Pölten, Sankt Pölten
  - Medizinische Universität Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (4):
  - Imelda VZW , Gastro-Enterology, Bonheiden
  - Hôpital Erasme, Gastro-Enterology, Brussels
  - AZ Groeninge - Campus Sint-Niklaas, Kortrijk
  - H.-Hartziekenhuis Roeselare-Menen vzw, Roeselare
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BC Cancer Agency-Vancouver, Vancouver, British Columbia
  - The Royal Victoria Hospital-Barrie, Barrie, Ontario
  - Hopital du Sacre-Coeur, Montreal, Quebec
  - Centre Hospitalier de L'Universite de Montreal St-Luc, Montreal
  - Princess Margaret Hospital, Ontario
  - Hotel-Dieu de Quebec, Québec
- France (3):
  - Centre Regional de lutte contre le cancer Paul Papin, Angers
  - Hôpital Saint Antoine, Paris
  - Hôpital Beaujon, Paris
- Germany (6):
  - Kliniken Essen-Mitte, Essen
  - Klinikum Freising, Freising
  - Praxis für Innere Medizin, Dr. Oettle Helmut, Friedrichshafen
  - LMU Klinikum der Universität, Munich
  - Klinikum Oldenburg, Oldenburg
  - Universitätsklinikum Würzburg, Würzburg
- Italy (14):
  - I.R.C.C.S. "Giovanni Paolo II" - Istituto Oncologico, Bari
  - E. O. Ospedali Galliera, Struttura Complessa Oncologia Medica, Genova
  - Nazionale per la Ricerca sul Cancro, Genova
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Oncologia Medica Falck, Milan
  - Istituto Oncologico Veneto, Padua
  - IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero universitaria Pisana, Pisa
  - Arcispedale Santa Maria Nuova, Unità Operativa di Oncologia Medica, Reggio Emilia
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Istituto Nazionale Tumori "Regina Elena", Roma
  - Istituto Clinico Humanitas, Rozzano
  - Ospedale Casa Sollievo della Sofferenza IRCCS, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Russia (24):
  - Med Radiological Centre of the Russian Academy of Med Sciences, Obninsk, Kaluga Oblast
  - Tatarstan Republican Onc Ctr, Kazan', Tatarstan Republic
  - Altai Territorial Oncological Center, Barnaul
  - Chelyabinsk Regional Onc Ctr, Chelyabinsk
  - Ivanovo Regional Oncology Center, Ivanovo
  - Regional Oncological Center # 2, Magnitogorsk
  - Moscow City Clinical Hosp #57 Chemotherapy Dept, Moscow
  - Blokhin Cancer Research Center, Moscow
  - Russian Res Ctr of Radiology under the Fed Agency for Hi-Tech Med Care, Moscow
  - Russian Research Ctr of Surgery n.a. B.V. Petrovskiy under the Russian Academy of Med Sciences, Moscow
  - Central Clinical Hosp of the President of the Russian Federation, Moscow
  - Semashko Central Hosp #2, Moscow
  - Moscow Municipal Onc Hosp #62, Moscow Region
  - Omsk Regional Onc Ctr, Omsk
  - Orenburg Regional Onc Ctr, Orenburg
  - Pyatigorsk Affiliate of Stavropol Regional Onc Ctr, Pyatigorsk
  - Clinical Hosp # 122 n.a. L.G. Sokolov, Saint Petersburg
  - Leningrad Regional Clinical Hosp, Saint Petersburg
  - St. Petersburg State Med Academy n.a.Mechnikov, Saint Petersburg
  - Russian Research Ctr for Radiology and Surgical Technologies, Saint Petersburg
  - St. Petersburg City Onc Ctr, Saint Petersburg
  - Tula Regional Oncology Center, Tula
  - Bashkortostan Republican Onc Ctr, Ufa
  - Yaroslavl Regional Onc Ctr, Yaroslavl
- Spain (8):
  - Hospital Vall D´Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid
  - Hospital Virgen del Rocio, Seville
- Ukraine (12):
  - Dnepropetrovsk City Hosp #4, Dnipro, UK
  - Donetsk Regional Antitumor Ctr, Donetsk, UK
  - Kirovohrad Regional Oncology Center, Department of Chemotherapy, Kirovohrad, UK
  - National Institute of Cancer, Department of Tumors of Abdominal Cavity and Retroperitoneum, Kyiv, UK
  - Kyiv City Clinical Hospital #10, Center for Hepatic, Bile Duct and Pancreatic Surgery, Kyiv, UK
  - Volyn Regional Oncology Center Department of Oncochemotherapy, Lutsk, UK
  - Lviv Regional Diagnostics and Treatment and Diagnostics Onc Ctr, Lviv, UK
  - O.F. Herbachevskyi Regional Clinical Hospital, Surgery Center, Zhytomyr, UK
  - Kharkov Regional Onc Ctr, Kharkiv
  - Kherson Regional Onc Ctr, Kherson
  - Odessa Regional Onc Ctr, Odesa
  - Zaporizhia Medical Academy of Postgraduate Education, Zaporizhia

REFERENCES:
- [Background] Tabernero J, Chiorean EG, Infante JR, Hingorani SR, Ganju V, Weekes C, Scheithauer W, Ramanathan RK, Goldstein D, Penenberg DN, Romano A, Ferrara S, Von Hoff DD. Prognostic factors of survival in a randomized phase III trial (MPACT) of weekly nab-paclitaxel plus gemcitabine versus gemcitabine alone in patients with metastatic pancreatic cancer. Oncologist. 2015 Feb;20(2):143-50. doi: 10.1634/theoncologist.2014-0394. Epub 2015 Jan 12. PMID 25582141
- [Background] Chiorean EG, Von Hoff DD, Tabernero J, El-Maraghi R, Ma WW, Reni M, Harris M, Whorf R, Liu H, Li JS, Manax V, Romano A, Lu B, Goldstein D. Second-line therapy after nab-paclitaxel plus gemcitabine or after gemcitabine for patients with metastatic pancreatic cancer. Br J Cancer. 2016 Jul 12;115(2):188-94. doi: 10.1038/bjc.2016.185. Epub 2016 Jun 28. PMID 27351217
- [Background] Tehfe M, Dowden S, Kennecke H, El-Maraghi R, Lesperance B, Couture F, Letourneau R, Liu H, Romano A. nab-Paclitaxel Plus Gemcitabine Versus Gemcitabine in Patients with Metastatic Pancreatic Adenocarcinoma: Canadian Subgroup Analysis of the Phase 3 MPACT Trial. Adv Ther. 2016 May;33(5):747-59. doi: 10.1007/s12325-016-0327-4. Epub 2016 Apr 16. PMID 27085323
- [Background] Scheithauer W, Ramanathan RK, Moore M, Macarulla T, Goldstein D, Hammel P, Kunzmann V, Liu H, McGovern D, Romano A, Von Hoff DD. Dose modification and efficacy of nab-paclitaxel plus gemcitabine vs. gemcitabine for patients with metastatic pancreatic cancer: phase III MPACT trial. J Gastrointest Oncol. 2016 Jun;7(3):469-78. doi: 10.21037/jgo.2016.01.03. PMID 27284481
- [Background] Vogel A, Rommler-Zehrer J, Li JS, McGovern D, Romano A, Stahl M. Efficacy and safety profile of nab-paclitaxel plus gemcitabine in patients with metastatic pancreatic cancer treated to disease progression: a subanalysis from a phase 3 trial (MPACT). BMC Cancer. 2016 Oct 21;16(1):817. doi: 10.1186/s12885-016-2798-8. PMID 27769210
- [Background] Kunzmann V, Ramanathan RK, Goldstein D, Liu H, Ferrara S, Lu B, Renschler MF, Von Hoff DD. Tumor Reduction in Primary and Metastatic Pancreatic Cancer Lesions With nab-Paclitaxel and Gemcitabine: An Exploratory Analysis From a Phase 3 Study. Pancreas. 2017 Feb;46(2):203-208. doi: 10.1097/MPA.0000000000000742. PMID 27841795
- [Background] Tabernero J, Kunzmann V, Scheithauer W, Reni M, Shiansong Li J, Ferrara S, Djazouli K. nab-Paclitaxel plus gemcitabine for metastatic pancreatic cancer: a subgroup analysis of the Western European cohort of the MPACT trial. Onco Targets Ther. 2017 Feb 2;10:591-596. doi: 10.2147/OTT.S124097. eCollection 2017. PMID 28203092
- [Result] Ramanathan RK, Goldstein D, Korn RL, Arena F, Moore M, Siena S, Teixeira L, Tabernero J, Van Laethem JL, Liu H, McGovern D, Lu B, Von Hoff DD. Positron emission tomography response evaluation from a randomized phase III trial of weekly nab-paclitaxel plus gemcitabine versus gemcitabine alone for patients with metastatic adenocarcinoma of the pancreas. Ann Oncol. 2016 Apr;27(4):648-53. doi: 10.1093/annonc/mdw020. Epub 2016 Jan 22. PMID 26802153
- [Result] Chiorean EG, Von Hoff DD, Reni M, Arena FP, Infante JR, Bathini VG, Wood TE, Mainwaring PN, Muldoon RT, Clingan PR, Kunzmann V, Ramanathan RK, Tabernero J, Goldstein D, McGovern D, Lu B, Ko A. CA19-9 decrease at 8 weeks as a predictor of overall survival in a randomized phase III trial (MPACT) of weekly nab-paclitaxel plus gemcitabine versus gemcitabine alone in patients with metastatic pancreatic cancer. Ann Oncol. 2016 Apr;27(4):654-60. doi: 10.1093/annonc/mdw006. Epub 2016 Jan 22. PMID 26802160
- [Result] Goldstein D, Von Hoff DD, Moore M, Greeno E, Tortora G, Ramanathan RK, Macarulla T, Liu H, Pilot R, Ferrara S, Lu B. Development of peripheral neuropathy and its association with survival during treatment with nab-paclitaxel plus gemcitabine for patients with metastatic adenocarcinoma of the pancreas: A subset analysis from a randomised phase III trial (MPACT). Eur J Cancer. 2016 Jan;52:85-91. doi: 10.1016/j.ejca.2015.10.017. Epub 2015 Dec 1. PMID 26655559
- [Result] Portal A, Pernot S, Tougeron D, Arbaud C, Bidault AT, de la Fouchardiere C, Hammel P, Lecomte T, Dreanic J, Coriat R, Bachet JB, Dubreuil O, Marthey L, Dahan L, Tchoundjeu B, Locher C, Lepere C, Bonnetain F, Taieb J. Nab-paclitaxel plus gemcitabine for metastatic pancreatic adenocarcinoma after Folfirinox failure: an AGEO prospective multicentre cohort. Br J Cancer. 2015 Sep 29;113(7):989-95. doi: 10.1038/bjc.2015.328. Epub 2015 Sep 15. PMID 26372701
- [Result] Goldstein D, El-Maraghi RH, Hammel P, Heinemann V, Kunzmann V, Sastre J, Scheithauer W, Siena S, Tabernero J, Teixeira L, Tortora G, Van Laethem JL, Young R, Penenberg DN, Lu B, Romano A, Von Hoff DD. nab-Paclitaxel plus gemcitabine for metastatic pancreatic cancer: long-term survival from a phase III trial. J Natl Cancer Inst. 2015 Jan 31;107(2):dju413. doi: 10.1093/jnci/dju413. Print 2015 Feb. PMID 25638248
- [Result] Vogel A, Pelzer U, Salah-Eddin AB, Koster W. First-line nab-paclitaxel and gemcitabine in patients with metastatic pancreatic cancer from routine clinical practice. In Vivo. 2014 Nov-Dec;28(6):1135-40. PMID 25398812
- [Result] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Derived] Von Hoff DD, Cridebring D, Tian OY, Han H, Bhore R, Franco T, Ondovik MS, Louis CU. Analysis of the Role of Plasma 25-Hydroxyvitamin D Levels in Survival Outcomes in Patients from the Phase III MPACT Trial of Metastatic Pancreatic Cancer. Oncologist. 2021 Apr;26(4):e704-e709. doi: 10.1002/onco.13645. Epub 2021 Jan 11. PMID 33345430
- [Derived] McCleary-Wheeler AL, McWilliams R, Fernandez-Zapico ME. Aberrant signaling pathways in pancreatic cancer: a two compartment view. Mol Carcinog. 2012 Jan;51(1):25-39. doi: 10.1002/mc.20827. PMID 22162229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in a 1:1 ratio and the randomization was stratified by geographic region (Australia versus Eastern Europe versus Western Europe versus North America), Karnofsky performance status (70 to 80 versus 90 to 100), and by the presence of liver metastases (yes versus no)
Pre-assignment Details: 38 participants were randomized but not treated due to the participants request to withdraw after the randomization results became known. 1 participant was randomized to Gemcitabine and was treated with Albumin-bound paclitaxel ABI-007/Gemcitabine in error and analyzed as treated and included in the intent to treat population (ITT)
Groups:
- Albumin-bound Paclitaxel (ABI-007)/Gemcitabine (Gem): Albumin-bound paclitaxel (ABI-007)/Gemcitabine: ABI-007 125 mg/m^2 administered intravenously (IV) in combination with Gemcitabine 1000 mg/m^2 IV weekly for 3 weeks on Days 1, 8, and 15 followed by one week of rest
- Gemcitabine (Gem): Gemcitabine 1000 mg/m^2 administered IV weekly for 7 weeks through Day 43 followed by a week of rest (Cycle 1), followed by cycles of weekly administration for 3 weeks on Days 1, 8, and 15 followed by a week of rest (Cycle 2 onward)
Period: Overall Study
Arm/Group | Albumin-bound Paclitaxel (ABI-007)/Gemcitabine (Gem) | Gemcitabine (Gem)
Started | 431 (Started = Intent to Treat Population and includes all randomized participants) | 430 (Started = Intent to Treat Population and includes all randomized participants)
Treated Population | 421 (Treated population = all randomized patients who received at least one dose of study drug) | 402 (Treated population = all randomized patients who received at least one dose of study drug)
Completed | 26 (Completed = participants remaining on treatment at the time of the data cut off 17 Sept 2012) | 12 (Completed = participants remaining on treatment at the time of the data cut off 17 Sept 2012)
Not Completed | 405 | 418
Not completed — Progressive Disease | 196 | 245
Not completed — Adverse Event | 128 | 73
Not completed — Physician Decision | 25 | 18
Not completed — Protocol Violation | 10 | 6
Not completed — Withdrawal by Subject | 28 | 39
Not completed — Other | 7 | 10
Not completed — Withdrew prior to starting treatment | 11 | 27

BASELINE CHARACTERISTICS:
Population: For the Karnofsky Performance Status (KPS) baseline characteristic, some of the participants did not have a baseline KPS recorded by the clinical site.
Groups:
- Albumin-bound Paclitaxel (ABI-007)/Gemcitabine: ABI-007 125 mg/m^2 administered in combination with gemcitabine 1000 mg/m^2 weekly for 3 weeks followed by one week of rest.
  Albumin-bound paclitaxel (ABI-007)/Gemcitabine : ABI-007 125 mg/m^2 administered in combination with Gemcitabine 1000 mg/m^2 weekly for 3 weeks, Days 1, 8, and 15 followed by one week of rest
- Gemcitabine: Gemcitabine, 1000 mg/m^2 administered weekly for 7 weeks followed by a week of rest (Cycle 1), followed by cycles of weekly administration for 3 weeks followed by a week of rest (Cycle 2 onward).
  Gemcitabine : Gemcitabine, 1000 mg/m2 administered weekly for 7 weeks, Day 1 through Day 43 followed by a week of rest (Cycle 1), followed by cycles of weekly administration for 3 weeks, Days 1, 8, and 15 followed by a week of rest (Cycle 2 onward).
- Total: Total of all reporting groups
Arm/Group | Albumin-bound Paclitaxel (ABI-007)/Gemcitabine | Gemcitabine | Total
Number analyzed (Participants) | 431 | 430 | 861
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (10.70) | 63.0 (9.27) | 62.2 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 173 | 359
  Male | 245 | 257 | 502
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 9 | 17
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 16 | 16 | 32
  White | 378 | 375 | 753
  More than one race | 25 | 26 | 51
  Unknown or Not Reported | 3 | 4 | 7
Karnofsky Performance Status (KPS) [Number; unit: participants] — The Karnofsky Performance Status Scale (KPS) was designed to measure the level of participant activity and medical care requirements. A general measure of participant independence and has been widely used as a general assessment of participants with cancer. The Karnofsky score runs from 100 to 0, where 100 is "perfect" health and 0 is death. The primary purpose of its development was to allow physicians to evaluate a participant's ability to survive chemotherapy for cancer. Two participants from the Albumin bound paclitaxel arm and one from the Gemcitabine arm did not have KPS performed.
  participants
    100% = normal, no complaints, no signs of disease | 69 | 69 | 138
    90% = normal activity, few symptoms of disease | 179 | 199 | 378
    80% = normal activity, some symptoms of disease | 149 | 128 | 277
    70% = caring for self, unable to work | 30 | 33 | 63
    60% = needs help, can manage most tasks | 2 | 0 | 2
    50% = needs help often and medical care | 0 | 0 | 0
    40% = disabled; requires special care & assistance | 0 | 0 | 0
    30% = severely disabled; death is imminent | 0 | 0 | 0
    20% = hospitalized; requires supportive treatment | 0 | 0 | 0
    10% = Moribund, fatal processes progressing fast | 0 | 0 | 0
    0% = Dead | 0 | 0 | 0
Pancreatic Primary Tumor Location [Number; unit: participants] — Main location or area of the pancreas where the disease is detected at diagnosis. Unknown location refers to disease area not being specified.
  participants
    Head | 191 | 180 | 371
    Body | 132 | 136 | 268
    Tail | 105 | 110 | 215
    Unknown = not specified | 3 | 4 | 7
Number of Baseline Lesions (Target + Non-Target) [Number; unit: participants] — Target lesions are those measurable at baseline and are generally the largest lesions, most reliably measured and most representative of the participants sites of disease. Non target lesions are all of the sites of disease present at baseline not classified as target lesions. They include bone and cystic lesions and pleural/pericardial effusion/ascites. The Independent Radiology Reviewers (IRR) only evaluated scans for those with baseline and follow-up scans.
  participants
    1 | 1 | 0 | 1
    2 | 32 | 25 | 57
    3 | 7 | 7 | 14
    4 | 37 | 43 | 80
    5 | 8 | 8 | 16
    >5 | 276 | 262 | 538

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization to the date of death from all causes. Participants who did not die were censored at the last known time the participant was alive. Patient survival was summarized using Kaplan-Meier methods.
Time Frame: From randomization to death; until the data cut off 17 Sept 2012. The maximum time in follow up was 37 months.
Population: Intent to Treat population (ITT population) consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Albumin-bound Paclitaxel (ABI-007)/Gemcitabine: Albumin-bound paclitaxel (ABI-007)/Gemcitabine: ABI-007 125 mg/m^2 administered intravenously (IV) in combination with Gemcitabine 1000 mg/m^2 IV weekly for 3 weeks on Days 1, 8, and 15 followed by one week of rest
- Gemcitabine: Gemcitabine 1000 mg/m^2 administered IV weekly for 7 weeks through Day 43 followed by a week of rest (Cycle 1), followed by cycles of weekly administration for 3 weeks on Days 1, 8, and 15 followed by a week of rest (Cycle 2 onward)
Arm/Group | Albumin-bound Paclitaxel (ABI-007)/Gemcitabine | Gemcitabine
Number analyzed (Participants) | 431 | 430
months | 8.5 [7.89 to 9.53] | 6.7 [6.01 to 7.23]
Statistical Analysis 1: Comparison: Albumin-bound Paclitaxel (ABI-007)/Gemcitabine vs Gemcitabine; Test type: Superiority or Other; p < 0.0001, Stratified Log-rank Test — P-value was based on a stratified log-rank test stratified by randomization strata of geographic region (North America versus Others), Karnofsky performance score (70 to 80 versus 90 to 100), and presence of liver metastasis; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.617 to 0.835] — Hazard ratio of Albumin bound paclitaxel + gemcitabine/gemcitabine alone. The associated hazard ratio and two-sided 95% confidence interval were estimated using a stratified Cox proportional hazard model

2. Secondary Outcome: Progression-free Survival (PFS) by Independent Radiological Review (IRR)
Description: Progression-free survival was defined as the time from the date of randomization to the date of disease progression, or death (any cause) on or prior to the clinical cutoff date, whichever occurred earlier. Participants who did not have disease progression or had not died were censored at the date of the last tumor assessment, on or prior to the clinical cutoff, and the patient was progression free. If a patient began a new anti-cancer treatment prior to documented disease progression (or death), the patient was censored at the date of last assessment when the patient was documented as progression free prior to the intervention. Patients with two or more consecutive missing response assessments prior to a visit with documented progression (or death) were censored at the last date of tumor assessment when the patient was documented to be progression free. PFS was summarized using Kaplan-Meier methods.
Time Frame: Randomization until disease progression or death from any cause; Until the data cut off of 17 Sept 2012. The maximum time in follow up was 37 months.
Population: Intent to Treat population (ITT population) consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Albumin-bound Paclitaxel (ABI-007)/Gemcitabine | Gemcitabine
Number analyzed (Participants) | 431 | 430
months | 5.5 [4.47 to 5.95] | 3.7 [3.61 to 4.04]
Statistical Analysis 1: Comparison: Albumin-bound Paclitaxel (ABI-007)/Gemcitabine vs Gemcitabine; Test type: Superiority or Other; p < 0.0001, Stratified Log-rank Test — P-value was based on a stratified log-rank test by randomization strata of geographic region (North America versus Others), Karnofsky performance score (70 to 80 versus 90 to 100), and presence of liver metastasis (yes vs no); Hazard Ratio (HR) = .69, 95% CI 2-sided [0.581 to 0.821] — Hazard ratio of Albumin bound paclitaxel + gemcitabine / gemcitabine alone. The associated hazard ratio and two-sided 95% confidence interval were estimated using a stratified Cox proportional hazard model

3. Secondary Outcome: Percentage of Participants Who Achieved an Objective Confirmed Overall Response by Independent Radiological Review (IRR)
Description: Objective tumor response was summarized as the percentage of participants who achieved a confirmed complete (CR) or partial response (PR) based on an independent blinded radiology assessment of response using Response Evaluation Criteria in Solid Tumors (RECIST) guidelines. Using RECIST Version 1.0, participants were to achieve either a complete response (CR) defined as the disappearance of all known disease and no new sites or disease related symptoms confirmed at least 4 weeks after initial documentation or partial response (PR) defined as at least a 30% decrease in the sum of the longest diameters of target lesions and no progression in non-target lesions based on confirmed responses from the investigator assessment of best overall response during study treatment.
Time Frame: Assessment every 4 weeks after initial response; Day 1 to data cut off of 17 Sept 2013; maximum time on study 37 months
Population: Intent to Treat population (ITT population) consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Albumin-bound Paclitaxel (ABI-007)/Gemcitabine | Gemcitabine
Number analyzed (Participants) | 431 | 430
percentage of participants | 23 [19.1 to 27.2] | 7 [5.0 to 10.1]
Statistical Analysis 1: Comparison: Albumin-bound Paclitaxel (ABI-007)/Gemcitabine vs Gemcitabine; PA+G/PG = response rate ratio of albumin bound paclitaxel + gemcitabine / gemcitabine; Test type: Superiority or Other; p < 0.0001, Chi-squared; Response Rate Ratio = 3.19, 95% CI 2-sided [2.178 to 4.662] — Response rate ratio: albumin-bound paclitaxel + gemcitabine /gemcitabine alone

4. Other Pre Specified Outcome: Participants With Treatment Emergent Adverse Events (AE)
Description: A Treatment Emergent Adverse Event (TEAE) is as any AE occurring or worsening on or after the first treatment of any study drug, and within 30 days after the last dose of the last study drug. Severity grades according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE) on a 1-5 scale: Grade 1= Mild AE, Grade 2= Moderate AE, Grade 3= Severe AE, Grade 4= Life-threatening or disabling AE, Grade 5=Death related to AE.
Time Frame: Study drug initiation through 30 days after the last dose of study drug or EOS, whichever is later; Up to 696 days
Population: Treated patient population
Measure: Number; unit: participants
Arm/Group | Albumin-bound Paclitaxel (ABI-007)/Gemcitabine | Gemcitabine
Number analyzed (Participants) | 421 | 402
participants
  At least 1 AE | 417 | 395
  ≥ 1 Treatment related AE (TEAE) | 403 | 371
  At least 1 Serious Adverse Event (SAE) | 212 | 172
  ≥ 1 treatment related SAE | 121 | 53
  ≥ 1 Grade (GR) 3/4 AE | 370 | 298
  ≥ 1 Grade 3 or higher AE | 374 | 303
  ≥ 1 AE leading to stopping treatment | 149 | 95
  ≥ 1 AE leading to death | 18 | 18
  ≥ 1 AE leading to dose reduction of ABI-007 or Gem | 209 | 125
  ≥ 1 AE related dose interruption of ABI-007 or Gem | 11 | 10
  ≥ 1 AE related dose delay of ABI-007 or Gem | 276 | 192

5. Other Pre Specified Outcome: Number of Participants With Dose Reductions
Description: The number of participants with dose reductions occurring during the treatment period. Dose reductions are typically caused by clinically significant laboratory abnormalities and /or treatment emergent adverse events/toxicities.
Time Frame: Maximum time on treatment was 666 days
Population: Treated Population
Measure: Number; unit: participants
Arm/Group | Albumin-bound Paclitaxel (ABI-007)/Gemcitabine (Gem) | Gemcitabine (Gem)
Number analyzed (Participants) | 421 | 402
participants
  At least 1 alumbin bound paclitaxel dose reduction | 172 | 0
  At least 1 Gemcitabine dose reduction | 198 | 132

6. Other Pre Specified Outcome: Number of Participants With Dose Interruptions
Description: The number of participants with dose interruptions experienced by participants that occurred during the treatment period. Dose interruptions are typically caused by clinically significant laboratory abnormalities and /or treatment emergent adverse events/toxicities.
Time Frame: Maximum time on treatment was 666 days
Population: Safety population, includes participants who received at least one study treatment
Measure: Number; unit: participants
Arm/Group | Albumin-bound Paclitaxel (ABI-007)/Gemcitabine | Gemcitabine
Number analyzed (Participants) | 421 | 402
participants
  ≥ 1 Albumin-bound paclitaxel dose interruption | 2 | 0
  At least 1 Gemcitabine dose interruption | 8 | 9

7. Other Pre Specified Outcome: Number of Participants With Dose Delays/Doses Not Given
Description: The number of dose delays or doses not given experienced by participants during the treatment period. Dose delays are typically caused by clinically significant laboratory abnormalities and /or treatment emergent adverse events/toxicities. Treatment delays of no longer than 21 days allowed participants to recover from acute toxicity, otherwise participants were discontinued from further treatment except in the event of peripheral neuropathy.
Time Frame: Up to 666 days
Population: Treated Population
Measure: Number; unit: number of dose delays
Arm/Group | Albumin-bound Paclitaxel (ABI-007)/Gemcitabine | Gemcitabine
Number analyzed (Participants) | 421 | 402
number of dose delays
  At least 1 ABI-007 dose delay/Not given | 300 | 0
  At least ≥ 1 Gem dose delay/Not given | 295 | 230

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days after the last dose (a maximum of 666 days)
Arm/Group | Albumin-bound Paclitaxel (ABI-007)/Gemcitabine | Gemcitabine
Serious Adverse Events (participants affected / at risk) | 212/421 | 172/402
Other Adverse Events (participants affected / at risk) | 412/421 | 392/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albumin-bound Paclitaxel (ABI-007)/Gemcitabine (N=421) | Gemcitabine (N=402)
Vomiting (Gastrointestinal disorders) | 18 | 12
Abdominal Pain (Gastrointestinal disorders) | 11 | 10
Nausea (Gastrointestinal disorders) | 11 | 8
Diarrhoea (Gastrointestinal disorders) | 9 | 3
Ascites (Gastrointestinal disorders) | 4 | 5
Intestinal obstruction (Gastrointestinal disorders) | 4 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 1
Duodenal Obstruction (Gastrointestinal disorders) | 3 | 2
Colitis (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Impaired gastric empyting (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatic cyst rupture (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Large Intestine perforation (Gastrointestinal disorders) | 0 | 1
Pancreatic haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Splenic artery aneurysm (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 17 | 11
Cellulitis (Infections and infestations) | 8 | 5
Urinary Tract Infection (Injury, poisoning and procedural complications) | 6 | 1
Sepsis (Infections and infestations) | 5 | 5
Septic Shock (Infections and infestations) | 4 | 5
Bacterial Sepsis (Infections and infestations) | 3 | 0
Lower Respiratory tract infection (Infections and infestations) | 3 | 2
Catheter site infection (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 1
Klebsiella bacteraemia (Infections and infestations) | 2 | 0
Liver Abscess (Infections and infestations) | 2 | 3
Neutropenic sepsis (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0
Oral Candidiasis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tooth Infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Biliary abscess (Infections and infestations) | 0 | 1
Breast cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 27 | 9
Oedema peripheral (General disorders) | 6 | 3
Asthenia (General disorders) | 3 | 5
Fatigue (General disorders) | 3 | 2
General physical health deterioration (General disorders) | 2 | 1
Chills (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 1
Pain (General disorders) | 1 | 2
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Device occlusion (General disorders) | 0 | 2
Face oedema (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 3
Non-cardiac chest pain (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13 | 20
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 2
Anaemia (Blood and lymphatic system disorders) | 9 | 2
Neutropenia (Blood and lymphatic system disorders) | 4 | 1
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Dehyration (Metabolism and nutrition disorders) | 20 | 12
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Pseudohyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 10 | 5
Bile duct obstruction (Hepatobiliary disorders) | 4 | 3
Jaundice (Hepatobiliary disorders) | 4 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 9 | 12
Capilary leak syndrome (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Labile hypertension (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 2
Hypovolaemic shock (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Venous stenosis (Vascular disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 2 | 2
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 5
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 2
Ataxia (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 3
Myocardial Infarction (Cardiac disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 3
Cardiogenic shock (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 2
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Biopolar I disorder (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 2 | 3
Renal failure acute (Renal and urinary disorders) | 2 | 4
Renal colic (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Liver Function test abnormal (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Haemoglobulin decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 6
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Perihepatic abscess (Infections and infestations) | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0
Generalized oedema (General disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 6
Jaundice cholestatic (Hepatobiliary disorders) | 4 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albumin-bound Paclitaxel (ABI-007)/Gemcitabine (N=421) | Gemcitabine (N=402)
Fatigue (General disorders) | 247 | 183
Oedema peripheral (General disorders) | 194 | 123
Pyrexia (General disorders) | 160 | 111
Asthenia (General disorders) | 77 | 51
Chills (General disorders) | 48 | 34
Mucosal inflammation (General disorders) | 42 | 16
Pain (General disorders) | 24 | 8
Nausea (Gastrointestinal disorders) | 223 | 189
Diarrhoea (Gastrointestinal disorders) | 182 | 94
Vomiting (Gastrointestinal disorders) | 145 | 107
Constipation (Gastrointestinal disorders) | 122 | 111
Abdominal Pain (Gastrointestinal disorders) | 92 | 87
Abdominal pain upper (Gastrointestinal disorders) | 42 | 28
Dyspepsia (Gastrointestinal disorders) | 34 | 28
Stomatitis (Gastrointestinal disorders) | 31 | 14
Abdominal distension (Gastrointestinal disorders) | 16 | 29
Ascites (Gastrointestinal disorders) | 15 | 26
Alopecia (Skin and subcutaneous tissue disorders) | 212 | 21
Rash (Skin and subcutaneous tissue disorders) | 117 | 39
Pruritis (Skin and subcutaneous tissue disorders) | 34 | 20
Dry Skin (Skin and subcutaneous tissue disorders) | 24 | 9
Erythema (Skin and subcutaneous tissue disorders) | 24 | 13
Anaemia (Blood and lymphatic system disorders) | 175 | 131
Neutropenia (Blood and lymphatic system disorders) | 172 | 122
Thrombocytopenia (Blood and lymphatic system disorders) | 127 | 115
Leukopenia (Blood and lymphatic system disorders) | 58 | 39
Neuropathy peripheral (Nervous system disorders) | 116 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 107 | 17
Dysgeusia (Nervous system disorders) | 68 | 33
Headache (Nervous system disorders) | 60 | 38
Dizziness (Nervous system disorders) | 47 | 34
Decreased appetite (Metabolism and nutrition disorders) | 149 | 104
Dehydration (Metabolism and nutrition disorders) | 75 | 33
Hypokalemia (Metabolism and nutrition disorders) | 50 | 28
Hypoalbuminaemia (Metabolism and nutrition disorders) | 25 | 18
Hyperglycaemia (Metabolism and nutrition disorders) | 22 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 72 | 30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 71 | 61
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 64 | 14
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 24 | 13
Urinary tract infection (Infections and infestations) | 37 | 14
Oral candidiasis (Infections and infestations) | 33 | 15
Cellulitis (Infections and infestations) | 25 | 16
Weight decreased (Investigations) | 57 | 47
Alanine aminotransferase increased (Investigations) | 45 | 36
Haemoglobin decreased (Investigations) | 41 | 29
Aspartate aminotransferase increased (Investigations) | 38 | 35
Platelet count decreased (Investigations) | 33 | 25
Neutrophil count decreased (Investigations) | 26 | 19
Blood alkaline phosphatase increased (Investigations) | 21 | 30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 48 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 44 | 15
Back Pain (Musculoskeletal and connective tissue disorders) | 41 | 40
Bone pain (Musculoskeletal and connective tissue disorders) | 24 | 8
Insomnia (Psychiatric disorders) | 64 | 46
Depression (Psychiatric disorders) | 50 | 24
Anxiety (Psychiatric disorders) | 35 | 43
Hypotension (Vascular disorders) | 38 | 26
Deep vein thrombosis (Vascular disorders) | 30 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship/contents of any publication is determined by site and provides sponsor a publication prior to submission. Sponsor has 60 days to review and avoid editorial changes but may request site delete confidential data. If publication contains patentable matter, site agrees to delay publication for 60 days. If study is part of multicenter protocol, site agrees not to independently publish. If multicenter publication is not forthcoming in 18 months after study end, site may proceed accordingly.